CLINICAL TRIAL: NCT00882323
Title: Reduced Toxicity Fludarabine, Cyclophosphamide Plus Thymoglobulin Conditioning Regimen for Unrelated Donor Transplantation in Severe Aplastic Anemia
Brief Title: Reduced Toxicity Fludarabine (Flu) + Cyclophosphamide (CPM) + Rabbit Antithymocyte Globulin (rATG) Conditioning Regimen for Unrelated Donor Transplantation in Severe Aplastic Anemia (SAA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Korean Society of Pediatric Hematology Oncology (Network)
Responsible Party: The Korean Society of Hematology, The Korean Society of Pediatric of Hematology Oncology
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSPHO-SCT 0802
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclophosphamide; fludarabine; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine (Experimental)
  Interventions: Drug: Cyclophosphamide, Fludarabine, Thymoglobulin

INTERVENTIONS:
Drug: Cyclophosphamide, Fludarabine, Thymoglobulin — cyclophosphamide (60 mg/kg once daily i.v. on days -8, -7)
  fludarabine (40 mg/m2 once daily i.v. on days -6, -5, -4, -3, -2)
  thymoglobulin (2.5 mg/kg once daily i.v. on days -4, -3, -2)

SUMMARY:
Anti-thymocyte globulin (ATG) has been used in severe aplastic anemia as a part of the conditioning regimen. Among the many kinds of ATG preparations, thymoglobulin had been found to be more effective in preventing graft versus host disease (GVHD) and rejection of organ transplants. As the fludarabine based conditioning regimens without total body irradiation have been reported to be promising for transplantation from alternative donors in SAA, thymoglobulin was added to fludarabine and cyclophosphamide conditioning to reduce GVHD and to allow good engraftment in unrelated donor transplantation. Our previous phase II study of fludarabine, cyclophosphamide plus thymoglobulin conditioning resulted in good engraftment (100%) and survival rate (74%). But grade III/IV toxicities occurred in 25% of patients and all events were treatment related mortalities. As cyclophosphamide is more toxic agent than fludarabine, we plan a new phase II study re; 'reduced toxicity fludarabine, cyclophosphamide plus thymoglobulin conditioning regimen for unrelated donor transplantation in severe aplastic anemia' by reducing dosage of cyclophosphamide and increasing dosage of fludarabine.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of severe aplastic anemia defined by any two or three peripheral blood criteria and either marrow criterion.

   * Peripheral blood

     1. Neutrophils < 0.5 x 109/l
     2. Platelets < 20 x 109/l
     3. Corrected reticulocytes < 1%
   * Bone marrow

     1. Severe hypocellularity (< 25%)
     2. Moderate hypocellularity (25-30%) with hematopoietic cells representing < 30% of residual cells
2. No prior hematopoietic stem cell transplantation.
3. Age: no limits.
4. Performance status: ECOG 0-2.
5. Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases:

   * Heart: a shortening fraction > 30% and ejection fraction > 45%.
   * Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper
   * Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
6. Patients must lack any active viral infections or active fungal infection.
7. Appropriate donor is available: Matched in 6/6 of A, B, DR loci.
8. Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Malignant or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.
4. Congenital aplastic anemia including Fanconi anemia.
5. Manipulated bone marrow.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate engraftment potential of reduced toxicity fludarabine, cyclophosphamide plus thymoglobulin conditioning regimen for unrelated bone marrow transplantation in severe aplastic anemia. | From Nov. 2008 to Oct. 2012

SECONDARY OUTCOMES:
To evaluate toxicities of reduced toxicity fludarabine, cyclophosphamide plus thymoglobulin conditioning regimen for UBMT/PBSCT in SAA. | From Nov. 2008 to Oct. 2012
To evaluate overall and EFS rate after UBMT/PBSCT. | From Nov. 2008 to Oct. 2012
To evaluate GVHD and immunologic recovery after UBMT/PBSCT. | From Nov. 2008 to Oct. 2012

CONTACTS AND LOCATIONS:
Overall Officials: Hyo seop Ahn, M.D, Ph. D, Principal Investigator — The Korean Society of Pediatric Hematology Oncology
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kang HJ, Shin HY, Park JE, Chung NG, Cho B, Kim HK, Kim SY, Lee YH, Lim YT, Yoo KH, Sung KW, Koo HH, Im HJ, Seo JJ, Park SK, Ahn HS; Korean Society of Pediatric Hematology-Oncology. Successful engraftment with fludarabine, cyclophosphamide, and thymoglobulin conditioning regimen in unrelated transplantation for severe aplastic anemia: A phase II prospective multicenter study. Biol Blood Marrow Transplant. 2010 Nov;16(11):1582-8. doi: 10.1016/j.bbmt.2010.05.010. Epub 2010 May 26. PMID 20685256